CLINICAL TRIAL: NCT06098261
Title: Bioequivalence Trial of Bilastine Tablets in Healthy Subjects in a Single-Center, Open, Randomized, Single-Dose, Double-Cycle, Double-Crossover Fasting State
Brief Title: Bioequivalence Study of Bilastine Tablets in Healthy Chinese Subjects
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Principal Investigator, Cao Yu, Director of Clinical Trials Center of Affiliated Hospital of Qingdao University, The Affiliated Hospital of Qingdao University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: H-BLSTP-T-B-2023-HBKS-01
Record Dates: First submitted 2023-10-19; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Healthy
MeSH Terms: interventions — bilastine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test (T)-Reference (R) (Experimental): In this trial, 40 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group A: Test (T)-Reference (R), The washout period (dosing interval) between doses will be at least 7 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T) Bilastine; Drug: Reference (R) Bilastine
- Reference (R)-Test (T) (Experimental): In this trial, 40 healthy subjects are planned to be enrolled in fasting. According to the randomization table, subjects will be randomly assigned to the Group B: Reference (R)-Test (T), The washout period (dosing interval) between doses will be at least 7 days. After fasting for at least 10 hours.
  Interventions: Drug: Test (T) Bilastine; Drug: Reference (R) Bilastine

INTERVENTIONS:
Drug: Test (T) Bilastine — Specification: Bilastine 20mg. Produced and supplied by Shandong Hubble Kisen Biological Technology Co., Ltd.
Drug: Reference (R) Bilastine — Specification: Bilastine 20mg. Produced by Menarini International Operations Luxembourg S.A.

SUMMARY:
Using a single-center, open, randomized, single-dose, double-cycle, double-crossover trial design method (washout period of 7 days), 40 screened and qualified healthy subjects were randomly divided into 2 groups, the T-R group and the R-T group, with 20 subjects in each group. The enrolled subjects entered the Phase I clinical research center 1 day prior to the first cycle of dosing, and fasted for 10 h or more prior to dosing. On the morning of the day of administration, 1 tablet of Bilastine (20 mg) developed by Shandong Hubble Kisen Biological Technology Co., Ltd. or 1 tablet of Bilastine (20 mg) licensed by Menarini International Operations Luxembourg S.A. were administered orally on an empty stomach.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully aware of the purpose, nature, methodology and possible adverse effects of the experiment, volunteer to be subjects, and sign an informed consent form prior to the start of all study procedures; 2. Healthy male or female subjects ≥18 years of age; 3. Weight ≥50.0kg for men and ≥45.0kg for women; 4. Body mass index (BMI) within the range of 19.0~26.0kg/m2 (including threshold values); 5. Vital signs examination, physical examination, clinical laboratory tests (blood tests, urine tests, blood biochemistry tests, coagulation tests, infectious disease screening, etc.), 12-lead electrocardiograms, which show normal results or are judged by the investigating physician to be abnormal but not clinically significant; 6. All subjects of childbearing potential (including the male subject's partner) who do not plan to have children and voluntarily use appropriate and effective contraception from the time of signing up to 6 months after the end of the trial, and who do not plan to donate sperm or eggs; 7. Able to communicate well with the researcher and understand and comply with the requirements of this study.

-

Exclusion Criteria:

1. Allergy, e.g., a known history of allergy to a substance, or a known history of allergy to Bilastine and its excipients, or a history of other allergic diseases (asthma, urticaria, eczematous dermatitis);
2. Those who develop an acute illness during the pre-study screening phase or prior to study drug administration;
3. Those with a history of the following diseases or chronic/severe medical conditions that the investigator believes are still clinically significant, including but not limited to cardiovascular, digestive, genitourinary, respiratory, hematologic, endocrine, immune, psychoneurologic, and skeletal systems;
4. especially those with gastrointestinal dysfunction, peptic ulcer, gastrointestinal diseases, and other conditions that may affect the absorption, distribution, metabolism, and excretion of medications;
5. Those with a history of QT prolongation and/or tip-twist ventricular tachycardia (including a history of congenital long QT syndrome);
6. Who have had surgery within 6 months prior to screening, or plan to have surgery during the study, or who have had or plan to have surgery that would interfere with the absorption, distribution, metabolism, or excretion of the drug;
7. Those who have been vaccinated within 4 weeks prior to the trial or who plan to receive any vaccine during the trial or within 1 week of the end of the study;
8. Those who have used any medications (including prescription, over-the-counter, herbal, nutraceuticals, and functional vitamins) within 2 weeks prior to screening;
9. Participation in another clinical trial with an investigational drug or medical device intervention within 3 months prior to screening;
10. Have received a blood transfusion or used blood products within 3 months prior to screening, or have a history of blood donation, or have lost more than 400milliliter of blood for other reasons, or plan to donate blood or blood components during the study or within 1 week of study completion;
11. Those who consumed an average of more than 14 units of alcohol per week (1 unit = 360milliliter of beer or 45milliliter of liquor at 40% alcohol by volume or 150milliliter of wine) in the past year, or who were unable to abstain from alcohol within 48 hours prior to study drug administration and or who are unable to abstain from alcohol during the trial, or who have an alcohol breath test result greater than 0.0 mg/100milliliter;
12. Those who smoked ≥5 cigarettes per day in the 3 months prior to screening or who were unable to stop using any tobacco-based products, including any nicotine-containing cessation products, within 48 hours prior to study dosing and for the duration of the trial;
13. History of substance abuse (including repeated, heavy non-medical use of all types of narcotic drugs and psychotropic substances) or drug use within 3 months prior to screening, or positive urine drug screens [including morphine, methamphetamine, ketamine, marijuana (tetrahydrocannabinolic acid), etc.] within 3 months prior to screening.(THC), etc.] are positive;
14. Use of any non-steroidal anti-inflammatory drug or any drug that interacts with bilastine (ketoconazole, erythromycin, cyclosporine, ritonavir or diltiazem, lorazepam, etc.) within 28 days prior to screening;
15. Poor vascular puncture conditions, inability to tolerate venipuncture or a history of needle and blood phobia;
16. Those who have difficulty in swallowing or have special dietary requirements and cannot accept a uniform diet and corresponding regulations;
17. Those who ingested or were unable to stop ingesting any caffeine-containing, alcoholic beverages (including chocolate, tea, coffee, cola, etc.), as well as grapefruit or grapefruit products, and foods that interfere with the metabolism of the drug, such as dragon fruit, mango, pomelo, oranges, etc., in the 48h prior to the administration of the drug or during the trial period;
18. Strenuous exercise within 1 week prior to screening, or inability to stop strenuous exercise during the test period;
19. Those who, in the opinion of the investigator, have factors that make participation in this trial inadvisable;
20. Use of oral contraceptives in the 30 days prior to the trial;
21. Use of long-acting estrogen or progestin injections or implants in the 6 months prior to the trial;
22. Women of childbearing age who have had unprotected sex with a partner in the 14 days prior to the test;
23. Pregnant or lactating women. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-11-21 (Estimated); Primary Completion 2023-12-03 (Estimated); Study Completion 2024-09-27 (Estimated)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 48 hours
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC0-t) | 48 hours
  Area under the drug concentration-time curve from time 0 to the last accurately measurable concentration at sample collection time t
Area under the plasma concentration versus time curve (AUC0-∞) | 48 hours
  Area Under the Plasma Drug Concentration-Time Curve from Time 0 to Infinite Time